CLINICAL TRIAL: NCT03479554
Title: China Antihypertensive Trial in Acute Ischemic Stroke II
Acronym: CATIS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Soochow University (Other)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Chair of Epidemiology, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1109725
Record Dates: First submitted 2018-03-09; First posted 2018-03-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Acute Ischemic Stroke
Keywords: antihypertensive treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Randomization will be conducted centrally at the SDCC. The randomization will be stratified by participating hospitals and use of antihypertensive medication. In each stratum, patients will be randomly assigned to the early antihypertensive treatment group or the delayed antihypertensive treatment group within each block. The block size will be random among 4, 6, and 8. The early BP lowering group will receive antihypertensive treatment immediately according to the study protocol, and the delayed BP lowering group will discontinue antihypertensive treatment for the first seven days after randomization.
  The randomization schedules will be generated using SAS PROC PLAN in SAS and will be concealed at the SDCC. When an eligible participant is ready for randomization, the site investigator/study coordinator will log-in to a password-protected website to obtain the randomization assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study physicians and nurses will not be masked to patients' randomization assignments because of the different time points for initiating BP treatment between the two randomization groups. The data on BP will also be unmasked because they are management tools for attaining the specific treatment targets. However, the study neurologists and nurses who conduct the neurological and functional assessments and collect clinical outcome data at the baseline and follow-up examinations will be masked to patients' assignments. The members of the Outcome Adjudication Committee will also be masked to patients' randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early antihypertensive treatment group (Experimental): BP-lowering treatment will start immediately after randomization in the early antihypertensive treatment group.
  Interventions: Other: Early antihypertensive treatment
- Delayed antihypertensive treatment group (Active Comparator): All home antihypertensive medications will be discontinued in the first seven days after randomization. Study participants will receive antihypertensive treatment on day eight after randomization.
  Interventions: Other: Delayed antihypertensive treatment

INTERVENTIONS:
Other: Early antihypertensive treatment — The CATIS 2 trial is designed to test BP reduction strategies-early antihypertensive treatment vs. delayed antihypertensive treatment-rather than test the efficacy of individual antihypertensive drugs. Several antihypertensive agents, including angiotensin-converting enzyme inhibitors, calcium channel blockers, and diuretics will be used in the trial.
  BP-lowering treatment will start immediately after randomization in the early antihypertensive treatment group. The target treatment goals are:
  * Step 1 (within 24 hours after randomization): To lower systolic BP by 10-20% with an average of 15% (but systolic BP not lower than 130 mmHg and diastolic BP not lower than 80 mmHg) within the first 24 hours after randomization based on the participant's admission BP levels.
  * Step 2 (within 7 days after randomization): To achieve systolic BP below 140 mmHg (but not lower than 120 mmHg) and diastolic BP below 90 mmHg (but not lower than 70 mmHg) and maintain this BP level afterward.
  Arms: Early antihypertensive treatment group
Other: Delayed antihypertensive treatment — All home antihypertensive medications will be discontinued in the first seven days after randomization. Study participants will receive antihypertensive treatment on day eight after randomization and will target systolic BP <140 mmHg (but not lower than 120 mmHg) and diastolic BP <90 mmHg (but not lower than 70 mmHg) in two weeks. A BP check-up visit will be conducted in two weeks. If BP treatment goal is not achieved, antihypertensive medication will be titrated or a new medication will be added.
  Arms: Delayed antihypertensive treatment group

SUMMARY:
The investigators propose to conduct a multicenter randomized trial to test the primary hypothesis of whether early antihypertensive treatment starting between the first 24-48 hours after the onset of an acute ischemic stroke will reduce the risk of composite case-fatality and major disability (modified Rankin Scale score ≥3) at three months compared to delayed antihypertensive treatment (starting on day 8 after stroke onset). In the proposed China Antihypertensive Trial in Acute Ischemic Stroke II (CATIS-2), the investigators will recruit 4,776 patients from 100 hospitals within the China-US Collaborative Stroke Clinical Trial Network. Eligibility criteria for the trial participants include age ≥40 years, acute ischemic stroke confirmed by CT/MRI, symptom onset between 24-48 hours, and average systolic blood pressure (BP) between 140-200 mmHg at randomization. Patients with extracranial or intracranial artery stenosis (≥70%) in both sides or the affected side, NIH Stroke Scale score of ≥21, Glasgow Coma Scale score <8, preceding moderate or severe dependency (modified Rankin scale score 3-5), revascularization, intravenous thrombolytic therapy or mechanical thrombectomy will be excluded. All eligible patients will discontinue their home antihypertensive medications. Patients admitted within 24 hours of symptom onset will require a reevaluation prior to randomization at 24 hours after stroke onset. After randomization, patients in the early treatment group will immediately receive antihypertensive treatment aimed at lowering average systolic BP by 10-20% within the first 24 hours and achieving an average BP <140/90 mmHg within seven days. Patients in the delayed treatment group will discontinue antihypertensive medications for the first seven days. After seven days, both groups will receive antihypertensive treatment with a BP goal of <140/90 mmHg. The primary study endpoint is a composite outcome of death and major disability at three months. The major secondary endpoint will be the first recurrent stroke (hemorrhagic or ischemic) over three-month follow-up after randomization. Other secondary endpoints include ordered 7-level categorical score of the modified Rankin Scale, all-cause mortality, and major vascular events at three months. The proposed study provides 85% statistical power to detect a 15% reduction in the composite outcome of death and major disability over three months at a significance level of 0.05 for a two-sided test. Based on experience from our previous trials, we assumed a 25% event rate of the primary study endpoint and potential loss to follow-up of 5% over three months. The CATIS-2 trial will provide important information for the development of clinical guidelines in the early management of BP among patients with acute ischemic stroke for reducing mortality and major disability.

DETAILED DESCRIPTION:
Stroke is the leading cause of death in China and the second leading cause of death in the world. In addition, stroke is the leading cause of long-term disability worldwide and a major financial burden to society. It is estimated that there are probably more than 3 million new strokes every year in China. In 2013, more than 1.9 million Chinese adults died from stroke, which represented an increase of 47.7% from 1.3 million in 1990.

Elevated blood pressure (BP) is common in the acute phase of ischemic stroke, occurring in ≥75% of all patients. The early BP increase following ischemic stroke often reflects uncontrolled chronic hypertension. In addition, the potential causes of this transient rise include disturbed cerebral autoregulation, damage or compression of brain regions that regulate BP, neuroendocrine disturbance, and non-specific mechanisms such as headache, urine retention, and psychological stress. Several clinical trials have tested the effects of immediate BP lowering on adverse clinical outcomes in patients with acute ischemic stroke and showed a neutral effect on death or dependency. The China Antihypertensive Trial in Acute Ischemic Stroke (CATIS) suggested a beneficial effect of BP lowering on death or major disability (odds ratio [OR] 0.73, 95% confidence interval [CI] 0.55-0.96, p=0.03) and recurrent stroke (OR 0.25, 95% CI 0.08-0.74, p=0.01) among patients with acute ischemic stroke who received antihypertensive treatment between 24-48 hours in a subgroup analysis. There are important knowledge gaps in BP management in acute ischemic stroke, such as when is the optimal time for initiation of antihypertensive treatment.

The investigators propose to conduct a multicenter randomized controlled trial to test the primary hypothesis of whether early antihypertensive treatment starting between the first 24-48 hours after the onset of an acute ischemic stroke will reduce the risk of composite case-fatality and major disability (modified Rankin scale score ≥3) at three months compared to delayed antihypertensive treatment (starting on day 8 after stroke onset). Patients with acute ischemic stroke will be randomly assigned within the first 24-48 hours after stroke onset to the early and delayed treatment groups. Patients in the early treatment group will immediately receive antihypertensive treatment aimed at lowering average systolic BP by 10-20% (with a mean reduction of 15%) within the first 24 hours, achieving an average systolic/diastolic BP <140/90 mmHg within seven days, and maintaining this level afterward. Patients in the delayed treatment group will discontinue antihypertensive medications for the first seven days. After then, both groups will receive antihypertensive treatment with an average systolic/diastolic BP goal of <140/90 mmHg. The primary study endpoint will be a composite outcome of death and major disability (modified Rankin Scale score ≥3) at three months after randomization. The major secondary endpoint will be the first recurrent stroke (hemorrhagic or ischemic) within three months. Other secondary endpoints include ordered 7-level categorical score of the modified Rankin Scale, all-cause mortality, and major vascular events at three months.

In the proposed China Antihypertensive Trial in Acute Ischemic Stroke II (CATIS-2), the investigators will recruit 4,776 patients (2,388 for each group) from 100 hospitals within the China Stroke Clinical Research Network. Eligibility criteria for the trial participants include age ≥40 years, acute ischemic stroke confirmed by computed tomography (CT) or magnetic resonance imaging (MRI), symptom onset between 24-48 hours, and an average systolic BP between 140-200 mmHg. The proposed study provides 85% statistical power to detect a 15% reduction in the primary study endpoint at three months at a significance level of 0.05 for a two-sided test. Based on experience from our previous CATIS trial, we assumed an event rate of 25% for the primary study outcome and potential loss to follow-up of 5% over three months. To achieve the CATIS-2 study objectives, we plan to:

1. Recruit and randomize 4,776 eligible patients (2,388 for each group) to the early antihypertensive treatment group or the delayed antihypertensive treatment group according to the study eligibility criteria;
2. Achieve and maintain target treatment goals for BP in the randomization groups;
3. Follow a study-wide strategy to encourage a standard of care based on clinical guidelines for the treatment of acute ischemic stroke other than BP for all participants;
4. Obtain follow-up data on clinical endpoints, neurological and functional status for each participant according to the study protocol; and
5. Estimate the effect of early antihypertensive treatment vs. delayed treatment on the primary and secondary endpoints according to intention-to-treat analysis and conduct predefined subgroup analyses.

The CATIS-2 study will provide important information for the development of clinical guidelines in the early management of BP among patients with acute ischemic stroke for reducing mortality and major disability.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥40 years
* Acute ischemic stroke confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) of the head
* Stroke onset within 24-48 hours*
* Systolic blood pressure between 140-200 mmHg and diastolic blood pressure between 80-120 mmHg

Exclusion Criteria:

* Hemorrhagic stroke confirmed by CT or MRI of the head
* CT or MRI-diagnosed vascular malformation, tumor, abscess, or other major non-ischemic brain disease (e.g., multiple sclerosis)
* Extracranial or intracranial artery stenosis (≥70%) in both sides or the affected side based on imagine study
* Stroke caused by arteritis, migraine, vasospasm, or substance abuse
* Severe stroke (NIHSS score of ≥21)
* Coma (Glasgow Coma Scale [GCS] score <8)
* Preceding moderate or severe dependency (modified Rankin scale [mRS] score 3-5)
* Planned or probable revascularization (any angioplasty or vascular surgery) within 3 months after screening
* Intravenous thrombolytic therapy (such as intravenous rtPA) or mechanical thrombectomy
* Severe heart failure (NY Heart Association class III and IV) or left ventricular ejection fraction <35%
* Myocardial infarction or unstable angina within past 3 months
* History of atrial fibrillation.
* History of aortic dissection
* History of all-cause dementia
* Difficult-to-control hypertension (systolic blood pressure ≥170 mmHg despite use of ≥4 antihypertensive medications for ≥6 months)
* Acute renal failure or dialysis or estimated glomerular filtration rate (eGFR) <20 ml/min/1.73 m2
* Any clinical conditions judged by the clinic team to likely limit the adherence to study procedures
* Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders
* Unable to participate in the follow-up examination (e.g., cannot travel to the participating hospital)
* Participation in another clinical trial within 30 days
* Pregnant, currently trying to become pregnant, or of child-bearing potential and not using birth control
* Failure to obtain informed consent from a participant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4810 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Composite outcome of death and major disability | At 3 months
  The primary endpoint for the CATIS-2 trial is a composite outcome of death and major disability (modified Rankin score ≥3) at 3 months.

SECONDARY OUTCOMES:
Recurrent stroke | At 3 months
  The first recurrent stroke event (hemorrhagic or ischemic) over three months of follow-up.
Modified Rankin Scale | At 3 months
  Ordered 7-level categorical score of the modified Rankin Scale
All-cause mortality | At 3 months
  Total mortality from all causes
Major vascular disease events | At 3 months
  Vascular deaths, non-fatal stroke, non-fatal myocardial infarction, coronary revascularization, hospitalized or treated angina, and hospitalized or treated congestive heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Principal Investigator — Tulane University; Yilong Wang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital; Liping Liu, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. Sharing IPD will require IRB approval from Tiantan Hospital and other participating institutes in China.

REFERENCES:
- [Derived] Zhong C, Wang M, Liu D, Wei Y, Wang M, Peng Y, Chen J, Pan Y, Xu T, Wang Y, He J, Wang Y, Zhang Y, Liu L, Xie X. Antihypertensive Treatments After Acute Ischemic Stroke: to Continue or Not? Hypertension. 2026 Feb;83(2):e25575. doi: 10.1161/HYPERTENSIONAHA.125.25575. Epub 2025 Dec 5. PMID 41347304
- [Derived] Xie X, Zhong C, Liu X, Pan Y, Wang A, Wei Y, Liu D, Xu T, Jiang Y, Wang M, Jing J, Meng X, Obst K, Chen CS, Wang D, Wang Y, Zhang Y, He J, Wang Y, Liu L. Early Versus Delayed Antihypertensive Treatment After Acute Ischemic Stroke by Hypertension History. Stroke. 2025 Mar;56(3):631-639. doi: 10.1161/STROKEAHA.124.049242. Epub 2025 Jan 14. PMID 39807580
- [Derived] Wei Y, Xie X, Pan Y, Wang M, Wang A, Liu D, Zhao Z, Nie X, Duan W, Liu X, Zhang Z, Liu J, Zheng L, Shen S, Zhong C, Xu T, Jiang Y, Jing J, Meng X, Obst K, Chen CS, Li H, Leng X, Wang D, Wang Y, Zhang Y, He J, Wang Y, Liu L. Early vs Delayed Antihypertensive Treatment in Acute Single Subcortical Infarction: A Secondary Analysis of the CATIS-2 Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2430820. doi: 10.1001/jamanetworkopen.2024.30820. PMID 39212990
- [Derived] Liu L, Xie X, Pan Y, Wang A, Wei Y, Liu J, Nie X, Liu D, Zhao Z, Wang P, Shen S, Zhong C, Xu T, Wang D, Wang GC, Song D, Ma Y, Zhao J, Jiang Y, Jing J, Meng X, Obst K, Chen CS, Wang D, Wang Y, Zhang Y, Wang Y, He J; CATIS-2 Investigators. Early versus delayed antihypertensive treatment in patients with acute ischaemic stroke: multicentre, open label, randomised, controlled trial. BMJ. 2023 Oct 9;383:e076448. doi: 10.1136/bmj-2023-076448. PMID 37813418
- [Derived] Liu L, Wang Y, Xie X, Liu D, Wang A, Wang P, Shen S, Zhong C, Wei Y, Xu T, Pan Y, Jiang Y, Meng X, Wang D, Zhang Y, He J, Wang Y. China Antihypertensive Trial in Acute Ischemic Stroke II (CATIS-2): rationale and design. Stroke Vasc Neurol. 2021 Jun;6(2):286-290. doi: 10.1136/svn-2020-000828. Epub 2021 Mar 16. PMID 33727409